CLINICAL TRIAL: NCT02284490
Title: High-dose Pemetrexed to Treat Lung Adenocarcinoma With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rongjie Tao (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Rongjie Tao, Neurosurgery, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI003; ShandongCHI (Registry Identifier: ShandongCHI)
Record Dates: First submitted 2014-10-10; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Brain Metastases
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Pemetrexed 900 mg/m² every 21 days until disease progression.
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — Administered intravenously at a dose of 900 mg/m2 every 21 days until disease progression.
  Other Names: pemetrexed disodium; Alimta

SUMMARY:
This phase II trial is studying how well pemetrexed disodium works in treating patients with Lung Adenocarcinoma With Brain Metastases

DETAILED DESCRIPTION:
* Determine the 6-month progression-free survival rate in patients with Lung Adenocarcinoma With Brain Metastases treated with pemetrexed disodium.
* Determine the time to progression in patients with Lung Adenocarcinoma With Brain Metastases treated with pemetrexed disodium.

Secondary

* Determine the radiographic response in patients with Lung Adenocarcinoma With Brain Metastases treated with pemetrexed disodium.
* Determine the time to response in patients treated with this drug.
* Determine the duration of response in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Collect safety data on patients with intracranial tumors treated with this drug.

OUTLINE: Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically. PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed brain metastases from lung adenocarcinoma.
* Measurable (greater than 1 cm in diameter) tumor by CT scan or MRI.
* ECOG (Eastern Cooperative Oncology Group) Performance status of 0-1.
* Measurable disease as defined by bidimensionally measurable lesions with clearly defined margins by CT scan or MRI.
* Biopsy is not required if radiographic imaging is consistent with brain metastases.
* Must have failed prior whole-brain radiotherapy.
* Patients with leptomeningeal metastases with or without brain metastases are eligible for therapy (may be diagnosed by MRI or cytology).
* Karnofsky performance score ≥ 60
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 mg/dL (transfusion allowed)
* SGOT/SGPT < 3.0 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Creatinine < 1.5 mg/dL
* Creatinine clearance > 45 mL/min
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study and for 3 months after completing study treatment
* Women who are pregnant or breast-feeding are not eligible for study treatment
* Negative pregnancy test
* Able to take steroids, vitamin B12, or folate
* No significant medical illnesses or infection that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy

Exclusion Criteria:

* Symptomatic brain metastasis
* Have received prior radiotherapy for brain metastasis
* Unable or unwilling to take folic acid, vitamin B12 supplementation or dexamethasone (or equivalent corticosteroid); or any other inability to comply with protocol or study related procedures.
* A prior malignancy other than NSCLC, except carcinoma in situ of the cervix or non-melanoma skin cancer, adequately treated low grade [Gleason score <6] localized prostate cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence
* Serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the investigator, would compromise the safety of the patient and his/her ability to complete study.
* Inability to discontinue administration of aspirin at a dose >1.3g/day or other non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam).
* Presence of fluid accumulations in third spaces, e.g., ascite or pleural effusion, which can be detected clinically (during physical examination), and which cannot be adequately controlled by drainage or other procedures prior to inclusion in the study.
* Peripheral neuropathy > CTC Grade 2
* Patient compliance or geographic distance precluding adequate follow up.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Determine the 6-month progression-free survival rate in patients with brain metastases from lung adenocarcinoma treated with pemetrexed disodium. | 1.5 years

SECONDARY OUTCOMES:
Determine the radiographic response in patients with brain metastases from lung adenocarcinoma treated with pemetrexed disodium. | 2 years
Determine the time to response in patients treated with this drug. | 2 years
Determine the duration of response in patients treated with this drug. | 2 years
Determine the overall survival of patients treated with this drug. | 2 years
Collect safety data on patients with brain metastases from lung adenocarcinoma treated with this drug. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

REFERENCES:
- [Result] Bailon O, Chouahnia K, Augier A, Bouillet T, Billot S, Coman I, Ursu R, Belin C, Zelek L, Des Guetz G, Levy C, Carpentier AF, Morere JF. Upfront association of carboplatin plus pemetrexed in patients with brain metastases of lung adenocarcinoma. Neuro Oncol. 2012 Apr;14(4):491-5. doi: 10.1093/neuonc/nos004. Epub 2012 Feb 22. PMID 22362813
- [Result] Ito S, Ogawa Y, Harada H, Yamaguchi T, Munakata K. [Long-term survival of patient with brain metastases from lung cancer treated by pemetrexed monotherapy]. Gan To Kagaku Ryoho. 2012 May;39(5):793-6. Japanese. PMID 22584333
- [Result] Dinglin XX, Huang Y, Liu H, Zeng YD, Hou X, Chen LK. Pemetrexed and cisplatin combination with concurrent whole brain radiotherapy in patients with brain metastases of lung adenocarcinoma: a single-arm phase II clinical trial. J Neurooncol. 2013 May;112(3):461-6. doi: 10.1007/s11060-013-1079-5. Epub 2013 Feb 19. PMID 23420398
- [Result] Zhuang H, Yuan Z, Wang J, Zhao L, Pang Q, Wang P. Phase II study of whole brain radiotherapy with or without erlotinib in patients with multiple brain metastases from lung adenocarcinoma. Drug Des Devel Ther. 2013 Oct 8;7:1179-86. doi: 10.2147/DDDT.S53011. eCollection 2013. PMID 24133369
- [Result] Yang H, Yang X, Zhang Y, Liu X, Deng Q, Zhao M, Xu X, He J. Erlotinib in combination with pemetrexed/cisplatin for leptomeningeal metastases and cerebrospinal fluid drug concentrations in lung adenocarcinoma patients after gefitinib faliure. Target Oncol. 2015 Mar;10(1):135-40. doi: 10.1007/s11523-014-0326-9. Epub 2014 Jul 2. PMID 24985049